CLINICAL TRIAL: NCT02676232
Title: DARWeb: an Online Psychosocial Intervention for Children With Recurrent Abdominal Pain and Their Families.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitat Oberta de Catalunya (Other)
Collaborators: Ministerio de Economía y Competitividad, Spain (Other Government)
Responsible Party: Principal Investigator, Rubén Nieto, Rubén Nieto Luna, PhD, Universitat Oberta de Catalunya
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R464E; PSI2013-42413-R (Other Grant/Funding Number: Ministerio de Economía y Competitividad)
Record Dates: First submitted 2016-01-28; First posted 2016-02-08 (Estimated); Last update posted 2019-04-24 (Actual); Status verified 2019-04

CONDITIONS: Abdominal Pain
Keywords: Online Intervention; Recurrent Abdominal Pain; Children
MeSH Terms: conditions — Abdominal Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention (Experimental): Participants in this arm will follow DARWeb: an online psychosocial intervention for children with recurrent abdominal pain and their parents. This is composed by 7 units for parents and 7 units for children, that have been developed from the cognitive-behavioral model, including setting goals, relaxation and distraction techniques, changing maladaptive thoughts and assertive communication training. The team under the program only contact with families for sending reminders and to answer potential technical problems or doubts
  Interventions: Behavioral: DARWeb
- Control (No Intervention): Participants allocated in this arm will not receive intervention. However, they will be invited to participate once the families allocated to the experimental group complete the program.

INTERVENTIONS:
Behavioral: DARWeb — Psychosocial Intervention from the cognitive-behavioral model, including different but related units for parents and children with recurrent abdominal pain.
  Arms: Intervention

SUMMARY:
Chronic and recurrent pain is a very important issue in the society, and its treatment is challenging.

In children, one of the most common pain problems is recurrent abdominal pain. This problem can affect up to 12% of the children population, and can interfere on daily activities of both children and parents. Recurrent abdominal pain in children is also associated with other health problems, and can be related to problems in adulthood. Unfortunately, the current health system does not have an effective treatment for these children and their families. This is why the investigators propose an online intervention, DARWeb, for people in this situation.

DARWeb provides an innovative solution using Information and Communication Technology to facilitate access. It is also innovative because it is directed towards secondary prevention, in contrast to the majority of current treatments available for pain problems that are focused in reducing the impact of pain when it is already severe. Thus, the objective of DARWeb is to provide information and teach strategies to children and their parents that help them to cope with pain and prevent pain interference in their daily lives (in the short, medium and long term).

With this project, the investigators plan, first, to create a new version of their treatment program (DARWeb V2) from the results of the pilot study. Second, the investigators will test the effects of DARWeb V2 through a randomized clinical trial with a large sample, and they will assess the short, medium and long term effects. In addition, the investigators want to study which of the variables that are addressed in their intervention are responsible for the potential changes observed.

The investigators expect that their treatment program will be effective to reduce pain in the short, medium and long term.

ELIGIBILITY:
Inclusion Criteria:

* 9 to 15 years
* Recurrent abdominal pain (abdominal pain at least once at month during a period of three months)
* Low level of disability

Exclusion Criteria:

* Identifiable organic cause.
* Disability preventing them to follow an online intervention.
* Not having a computer with Internet access.
* Not being able to read in Spanish language.

Ages: 9 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 61 (Actual)
Dates: Start 2014-09; Primary Completion 2019-03 (Actual); Study Completion 2019-03 (Actual)

PRIMARY OUTCOMES:
Pain Intensity | 2 weeks after intervention
  Assessed with the abdominal Pain Index
Pain Frequency | 2 weeks after intervention
  Assessed with the abdominal Pain Index
Pain Intensity | 6 months after the intervention
  Assessed with the abdominal Pain Index
Pain Intensity | 12 months after the intervention
  Assessed with the abdominal Pain Index
Pain Frequency | 6 months after the intervention
  Assessed with the abdominal Pain Index
Pain Frequency | 12 months after the intervention
  Assessed with the abdominal Pain Index

SECONDARY OUTCOMES:
Quality of life | 2 weeks after intervention; 6 and 12 months.
  Assessed with the Pediatric Quality of Life Inventory
Disability | 2 weeks after intervention; 6 and 12 months.
  Assessed with the Functional Disability Inventory
Depression | 2 weeks after intervention; 6 and 12 months.
  Assessed with the Children Depression Inventory.

CONTACTS AND LOCATIONS:
Overall Officials: Rubén Nieto, PhD, Principal Investigator — Universitat Oberta de Catalunya
Locations (1):
- Universitat Oberta de Catalunya, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Nieto R, Hernandez E, Boixados M, Huguet A, Beneitez I, McGrath P. Testing the Feasibility of DARWeb: An Online Intervention for Children With Functional Abdominal Pain and Their Parents. Clin J Pain. 2015 Jun;31(6):493-503. doi: 10.1097/AJP.0000000000000199. PMID 25551478
- See also: Research team website — http://psinet.uoc.edu/courses/darweb/?lang=en